CLINICAL TRIAL: NCT00336986
Title: An Open-label, Dose Escalation Safety and Tolerability Study of Recombinant Human Interleukin-21 (Phase 1) Followed by an Open-label Treatment Study (Phase 2a) in Patients With Stage IV Malignant Melanoma
Brief Title: Efficacy Study of IL-21 to Treat Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN028-1614
Record Dates: First submitted 2006-06-14; First posted 2006-06-15 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cancer; Malignant Melanoma
MeSH Terms: conditions — Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: recombinant interleukin-21

SUMMARY:
This trial is conducted in Oceania. A phase 2a study to assess the effect on tumor size. At least 14 to a maximum of 40 patients, who have not previously received treatment for their stage IV disease, will be treated for 6 weeks. IL-21 will be administered intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed surgically incurable metastatic melanoma
* Patients must have measurable disease
* ECOG performance status of 0 or 1
* Expected life expectancy at least 4 months

Exclusion Criteria:

* History of and signs/symptoms of uncontrolled brain metastases or edema.
* Previous treatment with chemotherapy or any biological anti-cancer drug (prior adjuvant therapy with interferon-alpha is permitted as long as treatment was completed at least six months prior to study entry.)
* Radiotherapy: Radiation therapy within 4 weeks prior to entering the study.
* Receipt of any investigational drug for treatment of metastatic melanoma prior to this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Tumor size assessed according to international criteria | After 8 weeks

SECONDARY OUTCOMES:
Serum levels of antibodies against recombinant human IL-21.
Markers of immunomodulation in blood.
Safety evaluation.
Time to progression.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR; 1452), Study Director — Novo Nordisk A/S
Locations (7):
- Australia (7):
  - Novo Nordisk Investigational Site, Box Hill
  - Novo Nordisk Investigational Site, East Melbourne
  - Novo Nordisk Investigational Site, Heidelberg
  - Novo Nordisk Investigational Site, Malvern
  - Novo Nordisk Investigational Site, Nedlands
  - Novo Nordisk Investigational Site, Parkville
  - Novo Nordisk Investigational Site, Westmead

REFERENCES:
- [Result] Coquet JM, Skak K, Davis ID, Smyth MJ, Godfrey DI. IL-21 Modulates Activation of NKT Cells in Patients with Stage IV Malignant Melanoma. Clin Transl Immunology. 2013 Oct 18;2(10):e6. doi: 10.1038/cti.2013.7. eCollection 2013 Oct. PMID 25505948
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com